CLINICAL TRIAL: NCT06632262
Title: An Open-label Phase 2, Multicenter, Open-Label Clinical Study to Evaluate the Safety and Efficacy of ABSK061 and ABSK043 with or Without Chemotherapy in Patients with Metastatic/Unresectable Solid Tumors with FGFR2/3 Alterations
Brief Title: A Phase 2 Clinical Study of ABSK061 and ABSK043
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSK061-201
Record Dates: First submitted 2024-10-01; First posted 2024-10-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: HER2-Gastric/Gastroesophageal Junction Cancer; Urothelial Carcinoma; Non-Small Cell Lung Cancer; Solid Tumors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): HER2-Gastric/Gastroesophageal Junction Cancer
  Interventions: Drug: ABSK061+ABSK043 in combination with CAPOX
- Cohort 2 (Experimental): Urothelial carcinoma
  Interventions: Drug: ABSK061 + ABSK043
- Cohort 3 (Experimental): Non-small cell lung cancer
  Interventions: Drug: ABSK061 + ABSK043
- Cohort 4 (Experimental): Other solid tumors
  Interventions: Drug: ABSK061 + ABSK043

INTERVENTIONS:
Drug: ABSK061 + ABSK043 — Participants with fibroblast growth factor receptor (FGFR) mutations and FGFR gene fusions will receive a dose of ABSK061 + ABSK043 oral capsule until disease progression, intolerable toxicity, withdrawal of consent, decision by the investigator to discontinue treatment, or end of data collection timepoint if there is clinical benefit in the opinion of the investigator, has been achieved.
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: ABSK061+ABSK043 in combination with CAPOX — Participants with HER2-Gastric/Gastroesophageal Junction Cancer and fibroblast growth factor receptor 2( FGFR2 ) amplification and overexpression will receive a dose of ABSK061 + ABSK043 oral capsule in combination with CAPOX until disease progression, intolerable toxicity, withdrawal of consent, decision by the investigator to discontinue treatment, or end of data collection timepoint if there is clinical benefit in the opinion of the investigator, has been achieved.
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity of ABSK061 + ABSK043 in terms of overall response rate (ORR) in in Patients with Metastatic/Unresectable Solid Tumors with FGFR2/3 Alterations

DETAILED DESCRIPTION:
ABSK061 is a selective and potent pan FGFR 2/3 inhibitor with demonstrated clinical activity in participants with a variety of FGFR inhibitors in a variety of solid tumors.

ABSK043 is a small molecule PD-L1 inhibitor with good oral bioavailability, high selectivity and high activity, and is currently being developed for the treatment of multiple cancers and potential non-oncology indications.

This study targets the underlying altered biology of FGFR-driven tumors irrespective of solid tumor histology subtype. The study consists of screening phase, treatment phase and the post treatment follow-up phase (from the end of treatment visit until the participant has died, withdraws consent, is lost to follow-up, or the end of study, whichever comes first). End of study is considered of the last visit of the last patient in this trial or the procedures shown in the schedule, or 12 months after the first dose of the last enrolled patient, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a measurable target lesion (per RECIST v1.1) (not applicable to expansion cohort 1) where:
* Dose Escalation: patients with histologically confirmed solid tumors who have progressed after standard of care, are unable to tolerate standard therapy, or have no standard of care currently available:
* Patients must have the a central laboratory or previous test report confirming FGFR2/3 gene activatingon alterations (including FGFR2/3 activating mutations, fusions/rearrangements, or FGFR2 amplifications) or overexpression in tumor tissue or blood based on central laboratory test or previous test reports.
* Expansion Phase:
* Cohort 1 (HER2-gastric/gastroesophageal junction cancer)
* Histologically or cytologically confirmed metastatic/unresectable gastric/gastroesophageal junction cancer, HER2 test negative
* The patient had FGFR2 amplification or overexpression in tumor tissue confirmed by a central laboratory test or a previous test report (previous test report only applied to FGFR2 amplification)
* Patients need to provide prior tumor tissue or willingness to undergo biopsy if no prior tumor tissue or insufficient quantity is required
* No prior (or up to one course of chemotherapy) systemic therapy for advanced gastric/gastroesophageal junction cancer, or disease progression more than 6 months after the end of the last prior adjuvant therapy
* Patients must have a measurable target lesion or evaluable non-target lesion (per RECIST v1.1)
* Cohort 2 (urothelial carcinoma)
* Histologically or cytologically confirmed metastatic/unresectable urothelial carcinoma with other histologic differentiation (including adenoid, squamous, or other types)
* Patients must have the prespecified a central laboratory or previous test report confirming the presence of a specific FGFR3 mutation or overexpression, FGFR2/3 fusion in tumor tissue or blood based on central laboratory test or previous test reports.
* No prior (or up to one course of chemotherapy) systemic therapy for advanced urothelial carcinoma, or disease progression more than 12 months after the end of the last prior adjuvant therapy, or disease progression or intolerable toxicity after at least one line of standard of care (per local standard of care or guidelines)
* Cohort 3 (non-small cell lung cancer)
* Histologically or cytologically confirmed metastatic/unresectable non-small cell lung cancer (NSCLC)
* Patients must have the prespecified a central laboratory or previous test report confirming the presence of a specific FGFR2/3 mutation, fusion, or overexpression in tumor tissue or blood based on central laboratory test or previous test reports.
* Disease progression or intolerable toxicity after at least one prior line of standard of care or targeted therapy for driver mutations (according to local standards of care or guidelines)
* Cohort 4 (Other Solid Tumors)
* Histologically or cytologically confirmed metastatic/unresectable other solid tumors
* Patients must have a central laboratory or previous test report confirmingthe FGFR2/3 gene activationng alterations (including FGFR2/3 activating mutations, fusions/rearrangements, or FGFR2 amplifications) or overexpression in tumor tissue or blood based on central laboratory test or previous test reports.
* Disease progression or intolerable toxicity after at least one prior line of standard therapy.

Exclusion Criteria:

* Previous treatment with an FGFR pathway inhibitor or a multi-kinase inhibitor designed to inhibit FGFR (consultation with the sponsor is recommended)
* Active or medical history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. (Patients with type 1 diabetes mellitus, hypothyroidism requiring hormone replacement therapy only, skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are allowed.Uncertain autoimmune-related status should be discussed with the sponsor).
* The patient had clinically symptomatic lung disease (e.g. interstitial pneumonia, pulmonary fibrosis, severe radiation pneumonitis, etc.) requiring systemic corticosteroid therapy within 6 months prior to enrollment.
* Known other malignancies that are in progression or require active treatment (except cured skin cancer, carcinoma in situ of the cervix, basal cell carcinoma, focal prostate cancer with a Gleason score of 6, focal prostate cancer with a Gleason score of 3 + 4 and treated for more than 6 months at screening).
* Time from the end of other prior anti-tumor therapy to the first dose of study drug: major surgery (palliative treatment for local lesions is allowed), in vitro and in vivo radiotherapy (> 30% bone marrow exposure) is less than 4 weeks; received immunotherapy or other antibody study drugs within 4 weeks prior to the start of study treatment; received chemotherapy (within 6 weeks of the start of study treatment with nitrosourea or mitomycin chemotherapy), endocrine therapy, and small molecule targeted therapy within 2 weeks or 5 half-lives, whichever is shorter.
* Patients who have not recovered to ≤ Grade 1 (CTCAE v5.0) from toxicities caused by prior chemotherapy, radiotherapy, and other anti-tumor therapies, including immunotherapy (except for alopecia as permitted by eligibility criteria or alopecia, vitiligo, stable hypothyroidism controlled by hormone replacement therapy, ≤ Grade 2 hearing loss, or ≤ Grade 2 peripheral neurotoxicity).
* History of ≥ Grade 3 immune-related adverse events with prior therapy.
* (Expansion Cohort 3 (non-small cell lung cancer)) Patients were previously identified with driver mutations (according to local diagnostic and therapeutic criteria or guidelines such as EGFR mutation, ALK rearrangement positive, KRAS G12C mutation positive, NTRK1/2/3 gene fusion positive, RET fusion positive, MET exon 14 skipping mutation, BRAF V600E mutation positive, ROS1 rearrangement positive) and did not receive targeted therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose limited toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Number of Participants With Adverse Event (AE), Serious Adverse Event, (SAE) and Laboratory Abnormalities Defined as Dose Limiting Toxicities (DLT)
To assess the tolerability of ABSK061 + ABSK043 in combination with CAPOX in patients with first-line gastric/gastroesophageal junction cancer | At the end of Cycle 1 (each cycle is 21 days)
  Number of Participants With Adverse Event (AE), Serious Adverse Event, (SAE) and Laboratory Abnormalities Defined as Dose Limiting Toxicities (DLT)
To assess the anti-tumor activity of ABSK061 + ABSK043 in combination with CAPOX as the primary endpoint of Progression-free survival (PFS) in first-line treatment of patients with metastatic/unresectable HER2-gastric/gastroesophageal junction cancer | up to 5 years
  PFS, as assessed by the investigator per RECIST v1.1
To assess the anti-tumor activity of ABSK061 + ABSK043 in patients with metastatic/unresectable urothelial cancer with FGFR2/3 activating alteration or FGFR3 overexpression, with Objective response rate (ORR) as the primary endpoint | up to 5 years
  Objective response rate (ORR): complete response and partial response determined by the investigator according to RECIST v1.1 and to be confirmed
To assess the anti-tumor activity of ABSK061 + ABSK043 in patients with non-small cell lung cancer withFGFR2/3 activating alteration or overexpression as the primary endpoint | up to 5 years
  PFS, as assessed by the investigator per RECIST v1.1
To assess the anti-tumor activity of ABSK061 + ABSK043 in patients with metastatic/unresectable other advanced solid tumors with FGFR2/3 activatingon alteration or overexpression as the primary endpoint | up to 5 years
  Objective response rate (ORR): complete response and partial response determined by the investigator according to RECIST v1.1 and to be confirmed

SECONDARY OUTCOMES:
Overall Response Rate as Assessed by Investigator | Up to 5 years
  Objective response rate (ORR): complete response and partial response determined by the investigator according to RECIST v1.1 and to be confirmed
Duration of Response (DOR) | Up to 5 years
  DOR is the duration from the date of initial documentation of a response to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study), or death, whichever comes first.
Disease Control Rate (DCR) | up to 5 years
  DCR is defined as the percentage of participants with CR, PR or stable disease (SD).DCR is defined as the percentage of participants with CR, PR or stable disease (SD).
Progression Free Survival (PFS) | up to 5 years
  PFS is the duration from the date of the first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death, whichever comes first.
Overall Survival (OS) | up to 5 years
  OS will be measured from the date of first dose of study drug to the date of the participant's death.
Maximum observed concentration(Cmax) | From date of enrollment #Day1# until the date of end of treatment visit, assessed up to 12 months
  To assess the PK profile of ABSK061 and ABSK043 after dosing of ABSK061 + ABSK043
Area under the concentration-time curve(AUC) | From date of enrollment #Day1# until the date of end of treatment visit, assessed up to 12 months
  To assess the PK profile of ABSK061 and ABSK043 after dosing of ABSK061 + ABSK043
Time to maximum observed concentration(Tmax) | From date of enrollment #Day1# until the date of end of treatment visit, assessed up to 12 months
  To assess the PK profile of ABSK061 and ABSK043 after dosing of ABSK061 + ABSK043

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Fudan University
Locations (21):
- China (21):
  - Guizhou Provincial People'S Hospital, Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Heibei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Central Hospital, Changsha, Hunan
  - Jiangxi Cance Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - ZhongShan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Xiangyang Central Hospital, Xiangyang, Sichuang
  - Changzhi People's Hospital, Changzhi
  - West China Hospital, Sichuan University, Chengdu
  - The First Hospital of China Medical University, Hangzhou
  - Zhejiang Provincial People'S Hospital, Hangzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - First Hospital of Shanxi Medical University, Xi'an
  - Shanxi Cancer hospital (Shanxi Cancer institute), Xi'an
  - First Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: Yes